CLINICAL TRIAL: NCT06685627
Title: Core Temperature in Open Water Wetsuited Swimming: a Cohort Study
Brief Title: Core Temperature in Open Water Wetsuited Swimming.
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other); Norwegian Armed Forces Medical Service (Other Government); SINTEF MiNaLab (Unknown)
Responsible Party: Principal Investigator, William James Morton, Principle Investigator, University Hospital, Akershus
Other Study IDs: Akershus Universitetssykehus
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Temperature
Keywords: Core temperature; water; swim; wetsuit; cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Open water wetsuited swimming. — All swimmers used their own well-fitting wetsuits (5 mm maximum thickness in accordance with World Triathlon guidelines7) and were free to supplement additional neoprene hats, gloves and booties as desired. A safety paramedic attended all swims. Swim distance was self-determined

SUMMARY:
Swimming in cold water is intrinsically unsafe. One of the threats is a fall in core body temperature (Tcore), which adversely affects all body systems and increases the risk of death. Wetsuits mitigate, but do not negate this threat. Environmental conditions may confound findings from laboratory studies or computer models, thus necessitating open water studies.

This study was designed to investigate the effects of open water wetsuited swimming on core body temperature at a range of different water temperatures between 8.4oC and 24.5oC.

ELIGIBILITY:
Inclusion Criteria:

* Trained and highly trained swimmers.

Exclusion Criteria:

* a history of cardiovascular disease, arrhythmias, or gastrointestinal abnormalities precluding the use of rectal temperature measurement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Trained and highly trained swimmers were recruited from local swim clubs and via social media
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2020-10-18 (Actual); Study Completion 2020-10-18 (Actual)

PRIMARY OUTCOMES:
Core temperature | The thermistor was inserted 15 minutes prior to immersion and measured the core temperature until 30 minutes after egress from the water.
  A self-inserted rectal pill was used to continuously measure core temperature in 76 open water swims by 31 wetsuited swimmers in water temperatures ranging from 8.4°C to 24.5°C. The Tcore curves were analysed by linear mixed model regression.

CONTACTS AND LOCATIONS:
Overall Officials: Jonny Hisdal, PhD, Study Director — Institute of Clinical Medicine, University of Oslo, Oslo, Norway
Locations (1):
- Institute of Clinical Medicine, University of Oslo, Oslo, Norway, Olso, Olso, Norway

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request from a validated body and subject to a data sharing agreement with the University of Oslo.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting data will be available from publication of the primary outcome data in a peer review journal and will be supported for 10 years form that date.
Access Criteria: IPD will be shared upon request from a validated body and subject to a data sharing agreement with the University of Oslo.

REFERENCES:
- [Derived] Morton WJ, Melau J, Olsen RA, Lovvik OM, Hisdal J, Sovik S. Thermal physiology of open water wetsuited swimming: A cohort study. Temperature (Austin). 2025 Mar 24;12(3):245-263. doi: 10.1080/23328940.2025.2479893. eCollection 2025. PMID 40926792